CLINICAL TRIAL: NCT06714747
Title: Soft Tissue Prediction in Orthognathic Surgery by Making Anatomically Accurate Virtual Model
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CH MAX FAC 21 01
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Orthognathic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of orthognathic surgery in the correction of dento-skeletal dysmorphies, whether they are Class II or Class III or asymmetries, is to improve both the function and aesthetic appearance of thepatient. Both aspects are equally important to achieve optimal results.

When the surgeon plans the surgery, he or she must therefore take into account the effects that bone displacements will have at the level of the soft tissues directly involved in the surgery, such as the maxilla and mandible. Traditionally, such surgery consists of an orthodontic presurgical phase1,2

.

DETAILED DESCRIPTION:
The role of orthognathic surgery in the correction of dento-skeletal dysmorphies, whether they are Class II or Class III or asymmetries, is to improve both the function and cosmetic appearance of the patient. Both aspects are equally important to achieve optimal results.

When the surgeon plans the surgery, he or she must therefore take into account the effects that bone displacements will have at the level of the soft tissues directly involved in the surgery, such as the maxilla and mandible. Traditionally, such surgery consists of an orthodontic presurgical phase1,2

.

The current knowledge of facial aesthetics and its changes consequent to orthognathic surgery is given by studies mainly carried out in 2-dimensions, performed using radiographs (teleradiographs of the skull in PA and LL) and standard photographic material, on which two-dimensional cephalometric and anthropometric studies have been performed. A first fragility, related to less realism, lies in the fact that these represent objects in 2-dimensions when the human body is a structure in 3-dimensions, as well as the chiurgy that is going to be performed and the resulting changes are in the 3-dimensions of space. A second lesser precision of this method of records acquisition is the substantial impossibility of obtaining comparable material in the preoperative and postoperative periods, due to the understandable difficulty of homogeneous acquisition of the records themselves: photographs and radiographs . Recent advances in technology have generated a wide variety of 3-D methods that allow acquisition in the 3-dimensions of space of both surface structures and skeletal bases. These methods include: digital stereophotogrammetry, CT, MRI, and ECO-3D.

This new knowledge has then enabled 3D studies that were previously done in 2D: cephalometry, morphological analysis of the face

. To date, commercially available simulation software manages to be fairly accurate with regard to hard tissues (bone, teeth), but not reliable enough with regard to simulation of soft tissues overlying skeletal bases and consensual motion in the face of facial hard tissue surgery, as they do not take into account the biomechanical variety of individual soft tissue components

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthognathic surgery and preoperative radiographic study with CBCT and MRI
* Patients with age > or = 18 years old
* Obtaining informed consent
* Patients with preoperative teleradiography and orthopantomography

Exclusion Criteria:

* patients with cleft lip-palate, facial malformations and/or syndromes (syndromes with involvement of the cephalic extremity, such as sd of Apert. Cropuzon, Ofeiffer, Treacher Collins)
* patients who have undergone application of Medpor prostheses or who have undergone ancillary procedures (lipofilling, fillers, volumetric facial augmentations with insertion of polyethylene ketone prostheses)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Verranno arruolati 10 pazienti retrospettivamente. Per ogni paziente verranno effettuate 27 simulazioni virtuali variando le proprietà biomeccaniche delle singole parti. I dati verranno perciò analizzati su 270 interventi virtuali. Le 27 simulazioni procapite vengono determinate in base al range di variazione che in fase iniziale si decide di dare ai vari parametri biomeccanici presi in considerazione per ogni componente del modello (tessuti molli, muscoli, osso)14
  .
  Un campione di 270 simulazione, consente di avere un intervallo di confidenza di 7.85 e un livello di confidenza del 99%. La tabella di seguito dimostra i valori massimi e minimi dati ai singoli muscoli per quanto riguarda il modulo di Young o modulo di elasticità.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
primary outcomes | 18 months
  Implementation of a virtual three-dimensional model of the face already provided for care procedure that is anatomically accurate in predicting soft tissue displacements following orthognathic surgery. This model will include the biomechanical characteristics of the facial muscles and skin.
  In particular, the sensitivities of different areas of the face (nose, cheeks, and upper lip) that are particularly important in orthognathic surgery will be evaluated in response to variation in the biomechanical properties of the muscles (Poisson's coefficient and Young's modulus).

SECONDARY OUTCOMES:
secondary outcomes | 18 months
  Demonstrate whether the inclusion of anatomical details such as facial muscles improves virtual prediction by comparing the simulation model with what is obtained in reality. This comparison will be made by superimposing the 3D object obtained from the virtual soft tissue simulation with the 3D soft tissue object obtained from postoperative CBCT. Through a colorimetric scale ranging from - to + 5 mm, we will evaluate the distance between the 3D reconstruction actually obtained from the patient's postoperative CBCT and the virtual simulation of the anatomically complex model.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Marchetti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS - Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna, Italy